CLINICAL TRIAL: NCT02777463
Title: The Prediction Using Diffusion-weighted MRI of the Response Evaluation in Borderline Resectable Pancreatic Cancer.
Brief Title: The Prediction Using Diffusion MRI of the Response Evaluation in BRPC in NAT.
Acronym: DIFFERENT
Status: Completed | Type: Observational
Sponsor: Wakayama Medical University (Other)
Responsible Party: Principal Investigator, Hiroki Yamaue, Second Department of Surgery, Wakayama Medical University, Wakayama Medical University
Other Study IDs: ADC-BRPC
Record Dates: First submitted 2016-05-11; First posted 2016-05-19 (Estimated); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: diffusion-weighted MRI — Diffusion MRI Patients undergo MRI within 3 weeks before start of neoadjuvant therapy/ 5 weeks after the last dose. The setting of MRI scans for b-values is 0, 50, 1000 s/mm2. The same MRI (the MRI system/scanner Intera Achieva 3.0T from Philips Medical Systems) in the independent institution is used for all patients analyzed on this study. The region of interest is determined by consensus between two experienced MR radiologists in a largest diameter based on images of abdominal CT scans avoiding the vascular area on the image of ADC map. The mean ADC values for each tumor are automatically calculated on the image of ADC map using a tomographic software program.

SUMMARY:
To investigate the correlation between pretreatment ADC value of diffusion MRI and pathologic response in patients with borderline resectable pancreatic carcinoma who undergo neoadjuvant therapy.

DETAILED DESCRIPTION:
Aim: The prediction using diffusion-weighted MRI of the response evaluation in borderline resectable pancreatic cancer.

Study design: Single institution. Single arm. Prospective Phase II Study.

Number of case: 28

Patients: The prediction using dMRI of the response evaluation in borderline resectable pancreatic carcinoma (BRPC) in neoadjuvant therapy.

Disease: Pancreatic carcinoma

Method: To investigate the correlation between pretreatment ADC value of diffusion MRI and pathologic response in patients with borderline resectable pancreatic carcinoma who undergo neoadjuvant therapy.

The correlation between pretreatment ADC value of diffusion MRI and pathologic response evaluated by Evans grade in patients with borderline resectable pancreatic carcinoma (BRPC) who undergo neoadjuvant therapy.

1. The correlation between pretreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction.
2. The correlation between posttreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction.
3. The correlation between the ratio of posttreatment/pretreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction.
4. The correlation between pretreatment ADC value of BRPC tumor in a largest diameter and the rate of tumor cell destruction.
5. The correlation between the ratio of posttreatment/pretreatment ADC value of BRPC tumor in a largest diameter and the rate of tumor cell destruction.
6. ADC Cut-off value which predict more than 50% and less than 10% in tumor cell destruction rate.
7. The correlation between the ratio of posttreatment/pretreatment ADC value of BRPC tumor in a largest diameter and the ratio of posttreatment/pretreatment SUV max.
8. ADC Cut-off value and SUV max cut-off value which predict survival time after surgery more than 2 years and less than 2 years.
9. The comparison of the accuracy of prediction for pathological diagnosis at abutment site between the ratio of posttreatment/pretreatment ADC value and CT scan.
10. Three correlation between high ADC value/low ADC value/the ratio of posttreatment/pretreatment ADC value and survival time after surgery.
11. Three correlation between high ADC value/low ADC value/the ratio of posttreatment/pretreatment ADC value and decreasing rate of CA19-9 value.
12. The correlation between tumor's limb sign in diffusion MRI and the rate of tumor cell destruction more than 10%.

ELIGIBILITY:
The patients with borderline resectable pancreatic cancer who is expexted to undergo neoadjuvant therapy and subsequent radical surgery.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The coefficient of correlation (Peason's r) was r=0.625 in our pilot study in patients with borderline resectable pancreatic cancer. To comfirm the producibility, it is judged as bad if the result is less than 10% from our previous study,the correlation coefficient threshold is 0.56 or more. At the setting of 90%confidential interval as 0.2, the number of case is estimated as 28. Considering unexpected situation, 30 cases is enough to analyze the correlation.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
The statistical analysis of the correlation between pretreatment ADC value of diffusion MRI and pathologic response evaluated by Evans grade in patients with borderline resectable pancreatic carcinoma (BRPC) who undergo neoadjuvant therapy. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.

SECONDARY OUTCOMES:
The statistical analysis of the correlation between pretreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between posttreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between the ratio of posttreatment/pretreatment ADC value at the abutment site of BRPC and the rate of tumor cell destruction. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between pretreatment ADC value of BRPC tumor in a largest diameter and the rate of tumor cell destruction. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between the ratio of posttreatment/pretreatment ADC value of BRPC tumor in a largest diameter and the rate of tumor cell destruction. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis by ROC curve to investigate ADC Cut-off value which predict more than 50% and less than 10% in tumor cell destruction rate. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between the ratio of posttreatment/pretreatment ADC value of BRPC tumor in a largest diameter and the ratio of posttreatment/pretreatment SUV max in PET-CT. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis by ROC curve to investigate ADC Cut-off value and SUV max cut-off value which predict survival time after surgery more than 2 years and less than 2 years. | Five years after initial therapy.
The statistical analysis of the comparison of the accuracy of prediction for pathological diagnosis at abutment site between the ratio of posttreatment/pretreatment ADC value and CT scan. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
Three correlation between high ADC value/low ADC value/the ratio of posttreatment/pretreatment ADC value and survival time after surgery. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between high ADC value/low ADC value/the ratio of posttreatment/pretreatment ADC value and decreasing rate of CA19-9 value. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.
The statistical analysis of the correlation between tumor's limb sign in diffusion MRI and the rate of tumor cell destruction more than 10%. | The time duration of examinations between pretreatment diffusion MRI and histopathological examination is approximately 4 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Wakayama Medical University, Wakayama, Wakayama, Japan